CLINICAL TRIAL: NCT03105453
Title: The Microbiome in Subfertility and Assisted Reproductive Technologies
Brief Title: The Microbiome in Subfertility and Assisted Reproductive Technologies (ART)
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, MD, PhD, Universitair Ziekenhuis Brussel
Other Study IDs: 2016/220
Record Dates: First submitted 2017-01-13; First posted 2017-04-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Infertility; Subfertility
Keywords: Assisted reproductive technologies; Microbiome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiome analysis using 16S ribosomal RNA sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study arm: Women in the study arm will undergo microbiome samplings described in the interventions section (3 sampling points)
  Interventions: Other: 3 Sampling points

INTERVENTIONS:
Other: 3 Sampling points — When entering the in-vitro fertilization/intracytoplasmatic sperm injection 4 samples will be harvested: a rectal swab, a cervical swab, a vaginal swab and an intra-uterine sample using an empty embryo catheter. After the ovarian stimulation treatment, the same patients will be sampled two more times: once at the moment of oocyte retrieval (rectal, cervical, vaginal and intra-uterine samples) and again just before the embryo transfer (at this stage, the embryo culture medium will be harvested, as well as an intra-uterine sample using the tip of an empty embryo inner catheter before the embryo transfer and a rectal sample)

SUMMARY:
To assess the impact of the female genital microbiome on ART outcome.

DETAILED DESCRIPTION:
The main objective of this study is to learn more about which microbial spectra are negatively or positively impacting IVF pregnancy outcome. This information is needed before proceeding to the next step in which an adaptation of the microbiome can be attempted to improve IVF outcome. The study is expected to shed light over the possible influence of the microbiome on causes for subfertility, endometrial receptivity and obstetrical complications. A diagnostic link may be found with entities that are often unexplained today, e.g. (recurrent) miscarriage and repeated implantation failure.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian women
2. Women undergoing an in-vitro fertilization cycle (for the first or second time)
3. Single embryo transfer
4. Day 5 embryo transfer
5. Gonadotropin-releasing hormone antagonist
6. Anti-mullerian hormone > 0,69 and < 3,5 µg/L
7. Body mass index ≤ 30 kg/m2
8. Signed informed consent

Exclusion Criteria:

1. Women suffering of chronic diseases which may impair pregnancy outcome (e.g. diabetes, chronic renal disease).
2. Antibiotics within 3 weeks of sampling
3. Surgical sperm retrieval
4. In-vitro maturation
5. Preimplantation genetic diagnosis
6. Grade 3 or 4 endometriosis
7. Patients unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing in-vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-09; Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 7 weeks
  To determine if there Is there a association between the microbiome profile and pregnancy outcome after ART

SECONDARY OUTCOMES:
Baseline microbiome profile | 1 week
  Descriptive analysis of the microbiome present in women suffering of infertility
Variation of microbiome profile during assisted reproductive technologies | 5 weeks
  Descriptive analysis of the microbiome present in women suffering of infertility according to the assisted reproductive technologies cycle stage
Microbiome profile of the embryo culture | 1 week
  Descriptive analysis of the microbiome present in the embryo culture on the day of embryo transfer
Live birth | 43 weeks
  To determine if there Is there a association between the microbiome profile and pregnancy outcome after assisted reproductive technologies

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, PhD, Study Director — Clinical head; Julie Bussche, Msc, Principal Investigator — Research collaborator
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Principal research site — http://www.brusselsivf.be/